CLINICAL TRIAL: NCT04861259
Title: A Phase III, Multicenter, Single-Arm Study Evaluating the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Crovalimab in Adult and Adolescent Patients With Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: A Study Evaluating the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Crovalimab in Adult and Adolescent Participants With Atypical Hemolytic Uremic Syndrome (aHUS)
Acronym: COMMUTE-a
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO42353; 2020-002475-35 (EudraCT Number); 2023-505089-27-00 (EU CTIS Number)
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atypical Hemolytic Uremic Syndrome
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Crovalimab (Experimental): Participants will be enrolled in three cohorts: [1] Naive Cohort - participants who have not been previously treated with complement inhibitor therapy; [2] Switch Cohort - participants who switch to crovalimab from another Complement Component 5 (C5) inhibitor and [3] C5 Single Nucleotide Polymorphism (C5 inhibitor) Cohort - participants with documented C5 polymorphism.
  Interventions: Drug: Crovalimab

INTERVENTIONS:
Drug: Crovalimab — Crovalimab will be administered at a dose of 1000 milligrams (mg) intravenous (IV) (for participants with body weight at least 40 (>=) and up to 100 kilograms (kg) or 1500 mg IV (for participants with body weight >=100kg) on Week 1 Day 1. On Week 1 Day 2 and on Weeks 2, 3 and 4, it will be administered at a dose of 340 mg subcutaneously (SC). On Week 5 and every 4 weeks (Q4W) thereafter, it will be administered at a dose of 680 mg SC (for participants with body weight >= 40kg to <100kg) or 1020 mg SC (for participants with body weight >=100kg).

SUMMARY:
This study aims to evaluate the efficacy and safety of crovalimab in adult and adolescent participants with aHUS.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >= 40 kg at screening.
* Vaccination against Neisseria meningitidis serotypes A, C, W, and Y; vaccination against serotypes B, according to national vaccination recommendations.
* Vaccination against Haemophilus influenzae type B and Streptococcus pneumoniae, according to national vaccination recommendations.
* For participants continuing to receive other therapies concomitantly with crovalimab (e.g., immunosuppressants, corticosteroids, mammalian target of rapamycin inhibitor (mTORi) , or calcineurin inhibitors): stable dose for >=28 days prior to screening and up to the first crovalimab administration.
* For female participants of childbearing potential: an agreement to remain abstinent or use contraception.
* Female participants of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of crovalimab.
* Participants with a prior kidney transplant are eligible if they have a known history of complement-mediated aHUS prior to the kidney transplant.
* Onset of initial TMA presentation within 28 days prior to the first dose of crovalimab (for Naive Cohort only).
* Documented treatment with either eculizumab or ravulizumab (for Switch Cohort only).
* Clinical evidence of response to a C5 inhibitor (for Switch Cohort only).
* Known C5 polymorphism (for C5 SNP Cohort only).
* Poorly controlled TMA following treatment with another C5 inhibitor (for C5 SNP Cohort only).

Exclusion Criteria:

* TMA associated with non-aHUS related renal disease.
* Positive direct Coombs test.
* Chronic dialysis within 90 days prior to first crovalimab administration and/or end stage renal disease.
* Identified drug exposure-related TMA.
* Presence or history of a condition that could trigger TMA, such as malignancy, bone marrow or organ transplant (other than kidney transplant) or autoimmune disease.
* History of a kidney disease, other than aHUS.
* History of Neisseria meningitidis infection within 6 months of study enrollment.
* Known or suspected immune deficiency (e.g., history of frequent recurrent infections).
* Positive Human Immunodeficiency Virus (HIV) test.
* Active systemic bacterial, viral, or fungal infection within 14 days before first crovalimab administration
* Presence of fever (>= 38°C)
* Multi-system organ dysfunction or failure.
* Recent intravenous immunoglobulin (IVIg) treatment.
* Pregnant or breastfeeding or intending to become pregnant.
* Participation in another interventional treatment study with an investigational agent or use of any experimental therapy within 28 days of screening or within five half lives of that investigational product, whichever is greater.
* Recent use of tranexamic acid.
* Current or previous treatment with a complement inhibitor (for Naive Cohort only).
* First initiation of plasma exchange/plasma infusions (PE/PI) should not be more than 28 days prior to first crovalimab administration (for Naive Cohort only).
* Last PE/PI completed less than 2 hours prior to first crovalimab administration (for Naive Chorot only).
* Receiving PE/PI within 8 weeks of the first crovalimab administration (Switch Cohort only).
* Positive for active Hepatitis B and C infection (HBV/HCV) (for Switch Cohort and C5 SNP Cohort participants who recently received C5 inhibitor treatment).
* Cryoglobulinemia at screening (for Switch Cohort and C5 SNP Cohort participants who recently received C5 inhibitor treatment).
* Diagnosis of condition leading to non-aHUS TMA: Thrombotic Thrombocytopenic Purpura (TTP), Shiga Toxin producing Escherichia Coli (STEC)
* TMA, Pneumococcal HUS, TMA secondary to cobalamin C defect and TMA related to a known DGKE nephropathy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2029-08-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Complete Thormbotic Microangiopathy Response (cTMAr) | Baseline up to Week 25 (after 24 weeks on treatment)

SECONDARY OUTCOMES:
Change from Baseline in Dialysis Status | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Change from Baseline in Chronic Kidney Disease (CKD) Stage | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Platelet Count | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Lactate Dehydrogenase (LDH) | Baseline up to Week 25 (after 24 weeks on treatment)
Observed Value in Hemoglobin | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Platelet Count | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Lactate Dehydrogenase (LDH) | Baseline up to Week 25 (after 24 weeks on treatment)
Change from Baseline in Hemoglobin | Baseline up to Week 25 (after 24 weeks on treatment)
Mean Change From Baseline in Fatigue (in Adult Participants only) | Baseline up to Week 25 (after 24 weeks on treatment)
  Assessed by the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Questionnaire.
  The FACIT-Fatigue (version 4) assesses self-reported fatigue and its impact upon daily activities and function. It consists of 13 items that assess fatigue using a 7-day recall period. Items are scored on a 0 (not at all) to 4 (very much) response scale. Relevant items are reverse scored and all items are summed to create total scores ranging from 0 [worse score] to 52 [better score].
Percentage of Participants with Platelet Count >= Lower Limits of Normal (LLN) (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Normalization of LDH (i.e. =< Upper Limit of Normal (ULN)) (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with >=25% Decrease in Serum Creatinine (Naive Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Time to cTMAr (Naive Cohort only) | Up to 8 years
Duration of cTMAr (Naive Cohort only) | Up to 8 years
Percentage of Participants with Ongoing cTMAr (Naive Cohort only) | At Week 25
Percentage of Participants with Maintained Thrombotic Microangiopathy Control (mTMAc) (Switch Cohort only) | Baseline up to Week 25 (after 24 weeks on treatment)
Percentage of Participants with Adverse Events (AEs) | Up to 8 years
Percentage of Participants with Injection-Site Reactions, Infusion-Related Reactions, Hypersensitivity, Malignant Hypertension (Including Malignant Renal Hypertension) and Infections (Including Meningococcal Meningitis) | Up to 8 years
Number of Participants with AEs Leading to Study Drug Discontinuation | Up to 8 years
Percentage of Participants with Clinical Manifestations of Drug-Target-Drug Complex (DTDC) Formation Amongst Those Participants who Switched to Crovalimab Treatment From Eculizumab Treatment or Ravulizumab Treatment | Up to Week 25
Serum Concentrations of Crovalimab Over Time | Up to 8 years
Prevalence of Anti-Crovalimab Antibodies at Baseline | Baseline
Percentage of Participants with Anti-Crovalimab Antibodies | Up to 8 years
Observed value of Pharmacodynamic Markers (CH50, Free/Total C5) | Up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- United States (7):
  - Univ of CA San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Emory Children's Center, Atlanta, Georgia
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - UT Health Science Center, San Antonio, Texas
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (3):
  - Santa Casa de Misericordia, Belo Horizonte, Minas Gerais
  - UPECLIN Hospital das Clinicas da Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Vancouver General Hospital, Vancouver, British Columbia, Canada
- Peking University First Hospital, Beijing, China
- France (4):
  - Hopital Lapeyronie, Montpellier
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Robert Debré, Paris
  - Hopital Tenon, Paris
- Germany (4):
  - Klinik II für Nephrologie, Rheumatologie, Diabetologie und Allgemeine Innere Medizin, Cologne
  - Universitätsklinikum Essen, Essen
  - Klinik für Nephrologie des Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
- Del- Pesti Centrumkorhaz- Szent Laszlo Korhaz Telephely, Budapest, Hungary
- India (2):
  - Medanta-The Medicity, Gurgaon, Haryana
  - All India Institute Of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
- Israel (3):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba MC, Ramat Gan
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
- Japan (3):
  - Nagoya University Hospital, Aichi
  - Saitama Medical University Hospital, Saitama
  - The University of Tokyo Hospital, Tokyo
- Mexico (4):
  - Hospital General de México, Distrito Federal, Mexico CITY (federal District)
  - Instituto Nacional de Ciencias, Mexico City, Mexico CITY (federal District)
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Hospital de Especialidades Puerta de Hierro S.A de C.V., Zapopan
- Instytut ?Centrum Zdrowia Matki Polki, Lodz, Poland
- Spain (2):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (4):
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Malatya Park Hospital, Malatya

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing